CLINICAL TRIAL: NCT01431131
Title: Ridge Preservation Comparing a Socket Allograft Alone to a Socket Allograft Plus a Facial Overlay Xenograft: A Clinical and Histologic Study In Humans
Brief Title: Ridge Preservation Comparing an Intrasocket Graft Alone to an Intrasocket Graft Plus a Facial Overlay Graft
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Henry Greenwell, Principal Investigator, University of Louisville
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 11.0352
Record Dates: First submitted 2011-09-07; First posted 2011-09-09 (Estimated); Results first posted 2017-01-31 (Estimated); Last update posted 2017-01-31 (Estimated); Status verified 2016-12

CONDITIONS: Clinical Efficacy
Keywords: graft placement; bone resorption
MeSH Terms: conditions — Bone Resorption

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intrasocket graft (Active Comparator): Positive control
  Interventions: Procedure: Intrasocket graft
- Intrasocket plus facial overlay graft (Experimental): Intrasocket cancellous allograft plus a facial overlay bovine xenograft
  Interventions: Procedure: Intrasocket plus facial overlay graft

INTERVENTIONS:
Procedure: Intrasocket graft — Intrasocket mineralized cancellous allograft
  Arms: Intrasocket graft
Procedure: Intrasocket plus facial overlay graft — Intrasocket mineralized cancellous allograft plus a facial overlay graft of bovine xenograft
  Arms: Intrasocket plus facial overlay graft

SUMMARY:
The purpose of this study is to compare two methods of ridge preservation in the maxillary anterior esthetic zone to determine the best method to establish adequate bone and soft tissue to accommodate implant placement. For the positive control group a mineralized cancellous allograft will be placed in the extraction socket. For the test group a mineralized cancellous allograft will be placed in the extraction socket plus an additional graft will be placed to overlay the facial surface of the socket that will be composed of bovine xenograft material. Outcomes will be clinical horizontal and vertical dimensional change and histologic analysis of the graft material at 4 months post-placement.

DETAILED DESCRIPTION:
Subjects met the eligibility criteria if they were at least 18 years of age and had one nonmolar tooth requiring extraction that would be replaced by a dental implant. Extraction sites were bordered by at least one tooth. Exclusion criteria included: 1) debilitating systemic diseases, or diseases that have a clinically significant effect on the periodontium; 2) molar extraction sites; 3) presence of or history of osteonecrosis of the jaws; 4) history of IV bisphosphonate treatment; 5) history of oral bisphosphonate treatment for more than three years; 6) pregnancy or lactation; 7) known allergy to any material or medication used in the study; 8) required antibiotic prophylaxis; 9) previous head and neck radiation therapy; 10) history of chemotherapy in the last 12 months; 11) long term steroid or non-steroidal anti-inflammatory drug therapy; or 12) failure to sign an informed consent approved by the Human Studies Committee. Patients were excluded post-treatment if they developed infection or had an adverse reaction to any of the materials used in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Have one non-molar tooth requiring extraction that will be replaced by a dental implant. The site must be bordered by at least one tooth.
2. Healthy person that is at least 18 years old.
3. Patients must sign an informed consent approved by the University of Louisville Human Studies Committee.

Exclusion Criteria:

1. Patients with debilitating systemic diseases, or diseases that have a clinically significant effect on the periodontium.
2. Molar teeth.
3. Presence of or history of osteonecrosis of the jaws.
4. Patients who are currently taking IV bisphosphonates or who had IV treatment with bisphosphonates irrespective of the duration.
5. Patients who have been treated with oral bisphosphonates for more than three years.
6. Pregnant women due to the possibility of miscarriage.
7. Patients with an allergy to any material or medication used in the study.
8. Patients who need prophylactic antibiotics.
9. Previous head and neck radiation therapy.
10. Chemotherapy in the previous 12 months.
11. Patients on long term NSAID or steroid therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-09; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Henry Greenwell, DMD, Principal Investigator — University of Louisville
Locations (1):
- Graduate Periodontics Clinic, School of Dentistry, University of Louisville, Louisville, Kentucky, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted between September 2011 and July 2012 in the Graduate Periodontics clinic at the University of Louisville School of Dentistry.
Groups:
- Intrasocket Graft: Positive control, an intrasocket cancellous allograft is placed
Period: Overall Study
Arm/Group | Intrasocket Graft | Intrasocket Plus Facial Overlay Graft
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Intrasocket Graft: Positive control, an intrasocket cancellous allograft was placed
- Total: Total of all reporting groups
Arm/Group | Intrasocket Graft | Intrasocket Plus Facial Overlay Graft | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 10 | 10 | 20
  >=65 years | 2 | 2 | 4
Age, Continuous [Mean (Standard Deviation); unit: years] | 52 (16) | 58 (11) | 55 (14)
Gender [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 4 | 7 | 11
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Horizontal Ridge Dimension
Description: WIll be measured with a digital caliper at baseline and 4 months.
Time Frame: Baseline and 4 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Intrasocket Graft | Intrasocket Plus Facial Overlay Graft
Number analyzed (Participants) | 12 | 11
mm | -1.6 (0.8) | -0.3 (0.9)

2. Secondary Outcome: Histologic Healing of the Osseous Graft
Description: Histologic analysis to determine vital bone, nonvital bone, and trabecular space percentages
Time Frame: 4 months
Measure: Mean (Standard Deviation); unit: percentage vital bone
Arm/Group | Intrasocket Graft | Intrasocket Plus Facial Overlay Graft
Number analyzed (Participants) | 12 | 11
percentage vital bone | 35 (16) | 40 (16)

ADVERSE EVENTS:
Time Frame: From the beginning to the end of the study.
Groups:
- Intrasocket Graft: Positive control, an intrasocket cancellous allograft will be placed
Arm/Group | Intrasocket Graft | Intrasocket Plus Facial Overlay Graft
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

LIMITATIONS AND CAVEATS:
There were no adverse events.

1 patient in the Intrasocket plus facial overlay graft group was excluded as an outlier. There was a large amount of bone gain and this skewed the data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No